CLINICAL TRIAL: NCT05381155
Title: tAckling intruSive Traumatic memoRies After chiLdbirth (ASTRAL): A Single-blind Waitlist Randomized Controlled Trial
Brief Title: Tackling Intrusive Traumatic Memories After Childbirth
Acronym: ASTRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antje Horsch, Associate professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-00652
Record Dates: First submitted 2022-05-13; First posted 2022-05-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder; Intrusive Traumatic Memories
Keywords: Posttraumatic Stress Disorder; Childbirth; Behavioral intervention; Randomized controlled trial; Visuospatial task
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single-blind waitlist randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in the immediate treatment group will receive the single-session behavioral intervention on day 15.
  Interventions: Behavioral: A single-session behavioral intervention composed of a brief evocation of the childbirth memory followed by a Tetris gameplay
- Waitlist (Other): Participants in the waitlist control group will receive the single-session behavioral intervention on day 30.
  Interventions: Behavioral: A single-session behavioral intervention composed of a brief evocation of the childbirth memory followed by a Tetris gameplay

INTERVENTIONS:
Behavioral: A single-session behavioral intervention composed of a brief evocation of the childbirth memory followed by a Tetris gameplay — The intervention is composed of two tasks:
  1. The childbirth narration task (8-10 min.): To trigger the malleability of the traumatic childbirth memory through memory reactivation, a psychologist will ask the participants to briefly narrate their childbirth and the moment associated with their most frequent or distressing CB-ITM. This intervention part will take place on the maternity ward to use this context as a reactivation cue.
  2. The visuospatial task (3 min. practice + 20 min. gameplay): Participants will be instructed to engage in a Tetris gameplay for 20 minutes on a handheld gaming device (Nintendo 3DS), which is assumed to disrupt memory reconsolidation. This part of the intervention will take place in a neutral room.

SUMMARY:
This single-blind waitlist randomized controlled trial aims to investigate the efficacy of a single-session behavioral intervention composed of a brief evocation of the childbirth memory followed by a visuospatial task (the computer game "Tetris"), on childbirth-related intrusive traumatic memories (CB-ITM) and other childbirth-related posttraumatic stress disorder (CB-PTSD) symptoms. Women who report CB-ITM after 6 weeks postpartum can be included in the study. Participants will be randomly allocated to either the immediate treatment (IT) group or to the waitlist (WL) group.

Women in the IT group will first report their CB-ITM in a daily diary during 2 weeks (diary 1). On the 15th day, they will meet a psychologist to receive the single-session behavioral intervention. They will then complete a daily diary during the 2 weeks post-intervention (diary 2) and during the 5th and 6th weeks post-intervention (diary 3).

Women in the WL group will report their CB-ITM continuously during 4 weeks in diary 1 and 2 before receiving the same intervention on the 30th day. They will also complete a last diary during the 2 weeks post-intervention (diary 3).

It is expected that women in the immediate treatment group (IT group) will have fewer CB-ITM in diary 2, in comparison to the WL group, for which we expect no significant change in the number of CB-ITM between diary 1 and 2.

This study will contribute to the development of a single-session behavioral intervention to reduce CB-ITMs and other CB-PTSD symptoms, which would reduce the distress experienced by mothers and may improve the well-being of the whole family.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Gave birth in one of the study centres
* Gave birth to a live baby
* Had at least 4 CB-ITM over the past two weeks
* Childbirth happened at least 6 weeks ago

Exclusion Criteria:

* Is not fluent enough in French to participate in the assessments
* Life-threatening illness of mother or infant
* Has an established intellectual disability or a psychotic illness
* Takes propranolol medication
* Alcohol and/or illicit drug abuse
* Is not able to distinguish ITM linked to other traumatic events from CB-ITM targeted during the intervention
* Has an ongoing psychological treatment in relation to her childbirth experience
* Is under 18 years old
* Being pregnant
* Perinatal loss of a child born during the index traumatic childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
The change in the number of maternal CB-ITM between the 2 weeks pre- and post-intervention | During the 2 weeks pre- and post-intervention
  The number of intrusive traumatic memories related to childbirth reported by participants in a diary during the 2 weeks pre- and post-intervention

SECONDARY OUTCOMES:
The change in the severity of maternal CB-PTSD symptoms between the 2nd week pre- and post-intervention | 2nd weeks pre- and post-intervention
  City Birth Trauma Scale (CiBTS)
The change in the number of maternal CB-ITM between the 2 weeks pre-intervention, and the 5th and 6th weeks post-intervention | During the 2 weeks pre-intervention, and the 5th and 6th weeks post-intervention
  The number of intrusive traumatic memories related to childbirth reported by participants in a diary during the 2 weeks pre-intervention, and during the 5th and 6th weeks post-intervention
The change in the severity of maternal CB-PTSD symptoms between the second week pre-intervention and the 6th week post-intervention | 2nd week pre- and 6th week post-intervention
  City Birth Trauma Scale (CiBTS)
The intervention acceptability assessed by participants from 30 to 60 days after the intervention | From 30 to 60 days after the intervention
  Acceptability questionnaire specifically designed for the study

OTHER OUTCOMES:
CB-ITM sensorial modalities, distress, nowness, and content | During 2-4 weeks pre-intervention, 2 weeks post-intervention, 5th and 6th weeks post-intervention
  Report of the sensorial modalities (visual, auditory, gustatory, olfactive, proprioceptive, tactile, and nociceptive) associated to the CB-ITM reported in the diary.
  Rating scale for psychological distress related to the CB-ITM that are reported in the diary on a scale ranging from 0 to 10 (0 = No distress at all while having the intrusion ; 10 = Extreme distress while having the intrusion).
  Rating scale of how much participants had the "impression that the memory was happening here and now" on a scale from 0 to 10 (0 = Not at all ; 10 = Extremely) while having the CB-ITM.
  Brief description of the content of the CB-ITM in the diary.
Participants' autonomic response and subjective distress during the intervention procedures | During the intervention procedures
  Autonomic response assessed via heart rate monitor during the intervention procedures.
  Rating scale for psychological distress assessed several times during the intervention using a Visual Analogue Scale of subjective distress going from 0 to 10 (0 = Not at all stressed and/or anxious ; 10 = Extremely stressed and/or anxious).
The change in postnatal depression and anxiety symptoms between the 1st week pre-intervention and the 6th week post-intervention | 1st week pre- and 6th week post-intervention
  Edinburgh Postnatal Depression Scale (EPDS) and Anxiety subscale of the Hospital Anxiety and Depression scale (HADS)
The change in the number of maternal CB-ITM between the 2 weeks post-intervention, and the 5th and 6th weeks post-intervention | During the 2 weeks post-intervention, and 5th and 6th weeks post-intervention
  The number of intrusive traumatic memories related to childbirth reported by participants in a diary during the 2 weeks post-intervention, and during the 5th and 6th weeks post-intervention
The change in the severity of maternal CB-PTSD symptoms between the 2nd week and 6th week post-intervention | 2nd and 6th weeks post-intervention
  City Birth Trauma Scale (CiBTS)

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, PhD, Principal Investigator — University of Lausanne and Lausanne University Hospital
Locations (2):
- Switzerland (2):
  - Maxime Haubry, Neuchâtel, Canton of Neuchâtel
  - Antje Horsch, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Yes
All IPD on which a publication is based will be shared in an anonymised form, at the time of the publication of the related outcomes, in an open access register.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available at the time of the publication of the related outcomes.
Access Criteria: Open access

REFERENCES:
- [Background] Horsch A, Vial Y, Favrod C, Harari MM, Blackwell SE, Watson P, Iyadurai L, Bonsall MB, Holmes EA. Reducing intrusive traumatic memories after emergency caesarean section: A proof-of-principle randomized controlled study. Behav Res Ther. 2017 Jul;94:36-47. doi: 10.1016/j.brat.2017.03.018. Epub 2017 Apr 6. PMID 28453969
- [Background] Deforges C, Fort D, Stuijfzand S, Holmes EA, Horsch A. Reducing childbirth-related intrusive memories and PTSD symptoms via a single-session behavioural intervention including a visuospatial task: A proof-of-principle study. J Affect Disord. 2022 Apr 15;303:64-73. doi: 10.1016/j.jad.2022.01.108. Epub 2022 Jan 30. PMID 35108604
- [Derived] Fort D, Deforges C, Messerli-Burgy N, Michael T, Baud D, Lalor J, Rimmele U, Horsch A. Tackling childbirth-related intrusive memories with a single-session behavioural intervention involving a visuospatial task: protocol for a single-blind, waitlist-controlled randomised trial. BMJ Open. 2023 May 29;13(5):e073874. doi: 10.1136/bmjopen-2023-073874. PMID 37247964